CLINICAL TRIAL: NCT05127252
Title: Impact of the Microbiome on Time to Pregnancy and Pregnancy Outcomes in Fertile Women Attempting to Conceive
Acronym: SweBioFertil
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Kenny Rodriguez-Wallberg, MD, PhD, Professor, Karolinska Institutet
Other Study IDs: Dnr 2021-03765
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Complications; Contraception; Pregnancy Loss; Fertility; Microbial Colonization; Metabolome
Keywords: cohort; fertility; microbiome; microbiota
MeSH Terms: conditions — Pregnancy Complications; Communicable Diseases | interventions — Metabolome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The samples will be analyzed on the high-throughput pipeline for microbiome studies at CTMR at KI. The pipeline includes standardized DNA extraction steps, library prep and shotgun metagenomic sequencing on the MGI sequencers available at the centre. Dedicated bioinformatic pipelines for taxonomy and functional capacity of the microbiome will be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vaginal and rectal microbiome and metabolome — Vaginal- and rectal sampling as a self-kit will be taken by the pat when ceasing the contraception at the midwife clinic when confirmed a clinical pregnancy and if a miscarriage occurs. If a miscarriage occurs additionally to the self-kit an endometrial biopsy will be taken.
  Other Names: SweBioFertil

SUMMARY:
This study aims to investigate the microbiome of women with previously proven fertility who plan to become pregnant.

DETAILED DESCRIPTION:
The women will be recruited at the time of removal of a copper or hormonal intrauterine device (IUD) or removal of a contraceptive implant at the barnmorskemottagningar (midwife clinics) in Stockholm's county in Sweden. A total of 500 women will be included in the study and will be followed until conception or up to the end of 1 year, whichever comes first. If conception occurs, the woman will be followed throughout pregnancy. Participant recruitment will take place over a period of two years.

ELIGIBILITY:
Inclusion Criteria:

* Women with a previous live birth in the past 5 years and planning a new pregnancy with the same male partner.
* 18-40 years of age
* Swedish personal identity number and a Swedish address (to send a sampling self-kit)
* Sufficient understanding of spoken and written Swedish or English to provide informed consent and complete the web-based questionnaire.

Exclusion Criteria:

* Women who do not have a child yet and plan to cease their contraception.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with previously proven fertility who plan to become pregnant. The women will be recruited at the time of removal of a copper or hormonal intrauterine device (IUD) or removal of a contraceptive implant
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The microbiome profile and metabolome associated with time to pregnancy, miscarriage, and live birth will be assessed. | 2024

SECONDARY OUTCOMES:
Microbiome profiles and metabolome related to obstetric outcomes | 2024
The microbiome profile for women above age >38 and women below <38. | 2024
The influence of BMI, medications and comorbidities on the microbiome profiles. | 2024
Microbiome profile for those women who don't conceive within a year. | 2024
The metabolome of the recognized microbiome for women with normal pregnancy outcomes | 2024
The metabolome of the recognized microbiome for women who develop miscarriage or other pregnancy complications | 2024

CONTACTS AND LOCATIONS:
Overall Officials: Lars Holmgren, Professor, Study Chair — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Reproductive Medicine, Karolinska University Hospital, Stockholm, Huddinge
  - Reproduktionscentrum Akademiska sjukhuset, Uppsala